CLINICAL TRIAL: NCT01861249
Title: A Multicenter Single-Arm Open Label Extension Study Evaluating The Long Term Safety And Tolerability Of SAR339658 In Patients With Ulcerative Colitis (UC)
Brief Title: Long Term Safety And Tolerability Of SAR339658 In Patients With Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was early terminated due to slow recruitment. Not linked to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS12593; 2013-001012-30 (EudraCT Number); U1111-1141-4634 (Other: UTN)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SAR339658 (Experimental): SAR339658, every 2 weeks (Q2W) or every 4 weeks (Q4W) according to clinical response at Week 8 in the ACT12688 trial
  Interventions: Drug: SAR339658

INTERVENTIONS:
Drug: SAR339658 — Pharmaceutical form: Solution for infusion
  Route of administration: Intravenous
  Other Names: Vatelizumab

SUMMARY:
Primary Objective:

To assess the long term safety and tolerability of SAR339658

Secondary Objective:

To assess the long term efficacy of SAR339658

DETAILED DESCRIPTION:
The study period per patient will include 62 weeks treatment, 6 weeks post treatment safety follow-up, followed by a long term safety follow-up performed in the form of a phone interview at 3, 6, 12, 18 and 24 months from the last administration of the study medication.

ELIGIBILITY:
Inclusion criteria:

* Patients with Ulcerative Colitis (UC) who were previously randomized and have completed the 8-week treatment in ACT12688 study with an acceptable safety profile. Patients who for administrative reasons could not be enrolled in the LTS12593 study right after completion of the 8-week treatment in the ACT12688 study must be enrolled within 3 months from the end of the ACT12688 study
* Signed written informed consent for Study LTS12593

Exclusion criteria:

* Patient with any adverse event leading to study drug (active or placebo) treatment discontinuation from ACT12688 study.
* Patient with any abnormalities or adverse events that per investigator judgment would adversely affect patient's participation in the long-term extension study.
* Use of any immunosuppressant (if patient is on immunosuppressant he or she must discontinue immunosuppressant before starting the LTS12593).
* If the patient started biological treatment for UC while waiting to be enrolled in the LTS12593, then he or she must stop the biological treatment and must have 8 weeks of wash out period before starting treatment with SAR339658 (only anti-tumor necrosis factors (TNFs) are allowed)
* Patients exposed to an anti-integrin or any investigational drug administered after the end of treatment in ACT12688
* Positive pregnancy test
* Breast feeding woman
* Women of childbearing potential not protected by highly effective contraceptive method of birth control and/or who are unwilling and unable to be tested for pregnancy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Events | Up to Week 68

SECONDARY OUTCOMES:
Percentage of participants with abnormal safety parameters (laboratory data and vital signs) | Up to Week 68
Proportion of participants with Clinical Remission by Mayo Score | At Week 62
Proportion of participants with Mucosal Healing | At Week 62
Change from baseline in the partial Mayo Score | At Weeks 10, 22, 34, 46 and 58
Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) | At Weeks 34 and 62

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (5):
  - Investigational Site Number 840059, Mission Hills, California
  - Investigational Site Number 840008, Miramar, Florida
  - Investigational Site Number 840048, Winter Park, Florida
  - Investigational Site Number 840024, Mexico, Missouri
  - Investigational Site Number 840088, San Antonio, Texas